CLINICAL TRIAL: NCT06818006
Title: Application of TAVI at Experienced Interventional Cardiac Centers Without On-site Cardiac Surgery
Brief Title: Application of TAVI at Experienced Interventional Cardiac Centers Without On-site Cardiac Surgery (ATLAS Study)
Acronym: ATLAS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATLAS-0000829-1
Record Dates: First submitted 2025-01-15; First posted 2025-02-10 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Aortic Stenosis; Severe Aortic Stenosis
Keywords: Aortic Stenosis; TAVR; TAVI; Sever aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: strategy study of two processes with path way of care
Who Masked: Outcomes Assessor
Masking Description: blinded clinical events adjudicated
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Active Comparator): EXPERIMENTAL ARM: TAVI WITHOUT ON-SITE SURGERY After randomization, the participant will be scheduled to undergo TAVI by experienced operators with appropriately trained cardiac catheterization staff.
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR) without surgical oversight
- Control Arms (Active Comparator): CONTROL ARM: TAVI WITH ON-SITE SURGERY After randomization, the patient will be scheduled to undergo TAVI by experienced operators with appropriately trained cardiac catheterization staff at an established TAVI center with on-site cardiac surgery
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR) with surgical oversight

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement (TAVR) with surgical oversight — Transcatheter Aortic Valve Replacement (TAVR) with surgical oversight
  Arms: Control Arms
Procedure: Transcatheter Aortic Valve Replacement (TAVR) without surgical oversight — Transcatheter Aortic Valve Replacement (TAVR) without surgical oversight
  Arms: Experimental Arm

SUMMARY:
The purpose of this study is to see if having the Transcatheter Aortic Valve Replacement (TAVR) procedure done in a hospital with onsite cardiac surgery available or not, makes a difference on participant outcomes. Current standard of care is to have this procedure done in a hospital with onsite cardiac surgery available.

Hypothesis

The investigators hypothesize that the TAVR in experienced interventional cardiac centers without on-site cardiac surgery will be safe and effective. Although this is happening clinically in select regions internationally, this change in the clinical application of TAVI requires a rigorous assessment of safety with a robust randomized trial and multicenter international collaboration.

DETAILED DESCRIPTION:
Primary Objectives:

The primary efficacy objective is to determine whether a Transcatheter Aortic Valve Implantation (TAVI) procedure performed by experienced operators in centers without on-site cardiac surgery is non-inferior to a TAVI procedure performed by experienced operators in centers with on-site cardiac surgery in terms of all-cause death, myocardial infarction, stroke and hospitalization for heart failure. The primary safety objective is to demonstrate that mortality associated with periprocedural complications actionable by emergent cardiac surgery (ECS) did not differ between study arms.

Research method/Procedures

ATLAS is an all-comer, prospective, randomized, multicenter, open label trial with blinded adjudicated evaluation of outcomes. The ATLAS study will involve centers without on-site cardiac surgery, but with experienced operators already performing TAVI. Participants will be recruited after Heart Team discussion and approval for TAVI. The eligibility of each participant will be confirmed by an established multidisciplinary Heart Team. Once approved for TAVI, dedicated review of the ATLAS study inclusion and exclusion criteria will occur. Study patients meeting inclusion and having no exclusion criteria will be randomized in a 2:1 fashion to TAVI performed in the experimental or standard of care arm stratified by two groups: 1) inoperable/high risk and 2) intermediate/low risk.

Randomization:

EXPERIMENTAL ARM: TAVI WITHOUT ON-SITE SURGERY After randomization, the participant will be scheduled to undergo TAVI by experienced operators with appropriately trained cardiac catheterization staff. CONTROL ARM: TAVI WITH ON-SITE SURGERY After randomization, the patient will be scheduled to undergo TAVI by experienced operators with appropriately trained cardiac catheterization staff at an established TAVI center with on-site cardiac surgery

Schedule of events:

1. Pre-eligibility screening 2. Inclusion/Exclusion criteria review 3. Randomization 4. 1-month post randomization 5. 3-months post randomization 6. TAVI procedure hospitalization 7. 1-month visit after TAVI 8. 12-month visit after TAVI 9. Final follow-up visit - 12-month post TAVI in control arm and equivalent median time post randomization in the intervention arm

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic AS reviewed and accepted for Transfemoral (TF) TAVI by an established Heart Team
* Obtained informed consent

Exclusion Criteria:

* Ambiguous aortic annular sizing on CT measurement deemed to increase the risk of valve embolization
* Hostile aortic root on CT for TAVI implantation defined by, but not limited to:
* High risk LVOT with a dimension significantly smaller than the annulus and/or extensive calcification
* Features that increase the risk of coronary artery occlusion including inadequate coronary artery height and/or shallow coronary sinuses in the setting of a significant coronary artery territory at risk (accounting for prior CABG)
* High risk STJ anatomy defined by inadequate height and/or diameter and/or excessive calcification
* Vascular anatomy with increased risk of ascending aorta trauma (i.e. combinations of existing ascending aortic aneurysm, and/or unfolded aorta and/or extensive tortuosity and/or excessive iliofemoral calcification)
* GFR <15, excluding patients on dialysis
* Life expectancy less than 3 years
* Any factor precluding 1-year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an Emergent CardiacSurgery (ECS) event: Ventricular | From enrolment to the end of 90 day follow up
  Primary Safety Outcome: Occurrence of an ECS event: Ventricular Valve Embolization, Aortic Annular Rupture, Ventricular Perforation requiring ECS or Ascending Aortic Dissection requiring ECS. Composite Endpoint of Primary Efficacy and Safety (Net clinical benefit)
  Multiple measurement will result in an outcome of ECS (Emergent Cardiac Surgery).
Death | From enrolment to the end of 90 day follow up
  Primary Efficacy Outcome: Composite of All Cause death from randomization.
Myocardial Infarction | From enrolment to the end of 90 day follow up
  Primary Efficacy Outcome: Composite of All Cause myocardial infarction (MI) from randomization.
Stroke | From enrolment to the end of 90 day follow up
  Primary Efficacy Outcome: Composite of All Cause Stroke, from randomization.
Heart Failure Hospitalization | From enrolment to the end of 90 day follow up
  Primary Efficacy Outcome: Composite of All Cause Heart Failure Hospitalization from randomization.

SECONDARY OUTCOMES:
Individual components of primary efficacy outcome | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Individual components of primary efficacy outcome
Hospitalization for cardiovascular cause | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Hospitalization for cardiovascular cause
Permanent Pace Maker (PPM) | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Need for Permanent Pace Maker (PPM) during study period
Urgent percutaneous coronary revascularization | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Need for urgent percutaneous coronary revascularization
Acute kidney injury | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Acute kidney injury requiring dialysis
Procedural wait time | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Procedural wait time from randomization to implantation date
Length of hospital stay | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Length of hospital stay (specific to TAVI implantation) hospitalization)
Total days of hospitalization | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Total days of hospitalization from randomization to end of study follow up
Health economics analysis- Adverse Events | From enrolment to the end of 90 day follow up
  Monitoring and analyzing of adverse events (AEs) weight and height will be combined to report BMI in kg/m^2).
Health economics analysis- Long-term Outcomes | From enrolment to the end of 90 day follow up
  Evaluation of the long-term effects of interventions on health and economic outcomes.
Health economics analysis- Healthcare Resource Utilization | From enrolment to the end of 90 day follow up
  Evaluation of the use of healthcare services, such as hospital admissions, outpatient visits, and medication usage.
Health economics analysis- Patient-Reported Outcomes (PROs | From enrolment to the end of 90 day follow up
  direct reports from patients about their health condition and treatment effects.
Quality of Life | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Quality of Life Baseline, 90 days post randomization, one year post randomization measured with Toronto Aortic Stenosis Quality of Life Questionnaire
Emergent balloon aortic valvuloplasty | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Need for emergent balloon aortic valvuloplasty prior to TAVI implantation required because of patent deterioration or emergent
Major Bleeding | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Major (type 2-4) bleeding (VARC). Multiple measurement to determine type of bleed.
Minor Bleeding | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Minor (type 1) bleeding (VARC). Multiple measurement to determine type of bleed.
Secondary Efficacy Outcomes | From enrolment to the end of 90 day follow up
  Secondary Efficacy Outcome: Major vascular complication (VARC)
  -Major or Minor vascular com
  Multiple measure to determine the vascular complications outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Mazankowski Heart Insitute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided